CLINICAL TRIAL: NCT02311270
Title: Survey on Cardiovascular Events in Patients With Metabolic Disease on Chronic Carnitine Supplementation
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: NAMDC7412
Record Dates: First submitted 2014-09-12; First posted 2014-12-08 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Metabolic Disorders
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about the effects of long term carnitine use in patients with metabolic disorders and its potential relationship to cardiovascular events.

DETAILED DESCRIPTION:
This online cross-sectional survey will examine the self-reported long-term carnitine use in patients with metabolic disorders and any potential relationship to cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mitochondrial disease or any other metabolic disorder
* Any age group
* NAMDC or RDCRN registry participant

Exclusion Criteria:

* Inability to provide informed consent and complete survey
* Lack of participation in NAMDC or RDCRN registry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients enrolled in the NAMDC portion of the RDCRN Contact Registry
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Assess how many patients with metabolic disorders are on chronic carnitine supplementation. | Up to one year from study activation.

SECONDARY OUTCOMES:
Assess how many patients who are on chronic carnitine supplementation have experienced a cardiovascular event. | Up to one year from study activation

CONTACTS AND LOCATIONS:
Overall Officials: Amel Karaa, MD, Study Chair — Massachusetts General Hospital
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- See also: Rare Diseases Clinical Research Network NAMDC page — http://www.rarediseasesnetwork.org/namdc